CLINICAL TRIAL: NCT01843959
Title: Abu Dhabi Diabetes and Obesity Study (ADOS) - A Study on the Aetiology and Associated Risk Factors of Patients With Obesity/Diabetes Within the Emirati Population.
Brief Title: Abu Dhabi Diabetes and Obesity Study
Status: Completed | Type: Observational
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Principal Investigator, Dr Nader Lessan, MD, Consultant Endocrinologist, Imperial College London Diabetes Centre
Other Study IDs: IREC008
Record Dates: First submitted 2013-04-25; First posted 2013-05-01 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Diabetes
Keywords: adenovirus-36; Emirati population
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Emirati Population: The individuals enrolled in this study will be divided into children (5-16 years of age) and adults (above 18). The groups will be further divided into BMI categories and glucose tolerance groups.
  * Group 1: Underweight (adjusted BMI <10th percentile) and no diabetes
  * Group 2:
  Normal weight (adjusted BMI 10th to 84.9th percentile) and no diabetes
  * Group 3:
  Overweight or obese children (adjusted BMI >= 85th percentile) and no diabetes
  * Group 4:
  Normal weight (adjusted BMI 10th to 84.9th percentile) and T1DM
  * Group 5:
  Overweight or obese children (adjusted BMI ≥ 85th percentile) and T1DM
  * Group 6:
  Normal weight (adjusted BMI 10th to 84.9th percentile) and T2DM
  * Group 7:
  Overweight or obese children (adjusted BMI ≥ 85th percentile) and T2DM

SUMMARY:
A cross-sectional study investigating the aetiology, mechanisms and associated complications contributing to obesity and diabetes within the UAE population. The study will be carried out in two main sample populations; children and adults, and characterized by the occurrence of obesity and diabetes. The main samples will then be divided into a subgroup for metabolomic analysis. Patients will be recruited from the Imperial College London Diabetes Centre. The study is aimed at elucidating the various factors that have an impact or may influence obesity and diabetes in the Emirati population.

DETAILED DESCRIPTION:
Obesity and Type 2 diabetes (T2DM) have been regarded as global epidemics in developed countries and more recently in developing nations. Obesity (a T2DM risk factor) and T2DM present significant health risks as individual diseases and substantial risks in individuals with both complications (Deepa Nath, 2006). The UAE and USA have a similar prevalence of obesity, 36% and 35.7% respectively. Interestingly, the percentage of the population with T2DM between the two groups differs significantly, 25% and 8.7% respectively. The rate of T2DM in the Emirati population is 2.9 fold higher than in the US. This suggests an altered inter relationship between obesity and T2DM. One hypothesis that could explain such a variation is differences in body metabolism and central adiposity between the two populations. This will be assessed by measuring cardiometabolic risk factors, central adiposity and metabolomics. Analysis of the metabolomic profiles may help define the risk factors associated with diabetes and differences in metabolic activity between various ethnicities.

Another area of ample interest is the advanced glycation end-products (AGEs) metabolic pathways (Pietropaoli D, 2012). AGEs are formed at an increased rate in diabetes and have a number of detrimental effects such as retinopathy, nephropathy and atherosclerosis (Melpomeni Peppa, 2003). As such, determining the core mechanisms that result in metabolic and cardiovascular dysfunction will aid in identifying and developing therapeutic targets, which may in turn alleviate the deleterious effects of respective disorders such as diabetes.

The aetiology of diabetes is complex. However, adenovirus 36 has been shown to play a significant role in obesity and diabetes. As such, analysis of ADV-36 occurrence within the Emirati population may provide insight into a novel obesity and diabetes risk factor and could further clarify the relationship between obesity and T2DM.

This study may provide evidence that clarifies how obesity can result in T2DM, and why this occurrence is more predominant in the Emirati population. In addition, the assessment of AGEs within the population, ranging from people with diabetes and obesity to healthy individual, may provide insight into potential therapeutic targets, thereby improving overall heath in the population. Finally, the data may improve our knowledge of new risk factors such as ADV-36 and their subsequent effects on diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All patients are eligible to participate in the study

Exclusion Criteria:

* Under 5 years of age

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Imperial College London Diabetes Centre, Abu Dhabi.
Sampling Method: Non-Probability Sample
Enrollment: 2130 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Percentage of the population in the U.A.E that are positive for adenovirus -36, specifically in children. | One year
  The initial aim of the study is to measure the prevalence of adenovirus 36 in the Emirati population.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Almgren M, Atkinson R, He J, Hilding A, Hagman E, Wolk A, Thorell A, Marcus C, Naslund E, Ostenson CG, Schalling M, Lavebratt C. Adenovirus-36 is associated with obesity in children and adults in Sweden as determined by rapid ELISA. PLoS One. 2012;7(7):e41652. doi: 10.1371/journal.pone.0041652. Epub 2012 Jul 27. PMID 22848557
- [Background] Atkinson RL. Adenovirus-36 and obesity. Pediatr Obes. 2012 Apr;7(2):e18-9. doi: 10.1111/j.2047-6310.2011.00043.x. No abstract available. PMID 22434760